CLINICAL TRIAL: NCT05555017
Title: Tracer-Based Image Guided Surgery for Recurrent Prostate Cancer: A Prospective Randomized Controlled Trial
Brief Title: Tracer-Guided Surgery for Recurrent Prostate Cancer
Acronym: Trace-II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N21TRA
Record Dates: First submitted 2022-09-15; First posted 2022-09-26 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: PSMA-radioguided surgery; ADT; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: ADT (Active Comparator): Patients in arm A will receive standard 6 months of ADT according to current clinical guidelines.
  Interventions: Drug: ADT
- Arm B: ADT + PSMA radioguided surgery (Experimental): Patients in arm B will receive standard 6 months of ADT according to current clinical guidelines, and will undergo 99mTechnetium (99mTc)-based PSMA-radioguided salvage surgery.
  Interventions: Procedure: PSMA-radioguided surgery; Drug: ADT

INTERVENTIONS:
Procedure: PSMA-radioguided surgery — Approximately 15-24 hours prior to surgery, 400-600 Megabecquerel (MBq) of 99mTc-PSMA-I&S will be intravenously administered to the patient at the Nuclear Medicine department. Following this injection patients will be allowed to return home, and then present for their 99mTechnetium (99mTc)-based PSMA-radioguided salvage surgery the next day.
  Arms: Arm B: ADT + PSMA radioguided surgery
Drug: ADT — Standard 6 months of ADT according to current clinical guidelines. ADT consists of one subcutaneous depot of 22,5mg triptorelin (Pamorelin), with 4 weeks bicalutamide 50mg per os from 2 weeks before till 2 weeks after the first Pamorelin administration.

SUMMARY:
ADT with or without robot-assisted PSMA-radioguided surgery for patients with recurrent prostate cancer.

DETAILED DESCRIPTION:
Improving the oncological treatment outcomes in men with a biochemical recurrence after primary prostate cancer (PC) treatment that are diagnosed with a disease recurrence confined to the regional lymph nodes or local residual disease using Prostate Specific Membrane Antigen (PSMA) Positron Emission Tomography and Computed Tomography (PET/CT.)

The proposed trial randomizes patients with recurrent PC following primary PC treatment to either 6 months of ADT or Technetium-PSMA-radioguided salvage surgery plus 6 months of ADT. Although the optimal duration of ADT is unknown, a minimal duration of 6 months of ADT seems advisable in this setting and will be mandatory for both arms.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged ≥ 18 years.
* Hormone-sensitive recurrent prostate cancer after radical prostatectomy, external beam radiotherapy or brachytherapy
* ≤ 2 lymph node metastases or local residual disease within the pelvis with sufficient PSMA expression (≥2 times regional vascular activity level) as determined by PSMA-based PET
* PSA-value < 4 ng/mL in case of a local recurrence and PSA < 3 ng/ml in case of (a) nodal recurrence(s)
* Had a PSMA PET/CT within 90 days before surgery
* Suitable for salvage surgery, as per institutional guidelines.
* Charlson Comorbidity Index ≤ 4
* World Health Organisation (WHO) performance status 0, 1, or 2.
* Written and signed informed consent.

Exclusion Criteria:

* Other diagnosis of malignancy or evidence of other malignancy within 5 years before screening for this study (except non-melanoma skin cancer).
* More than 2 lymph node metastases on PSMA PET/CT
* Suspicion of local recurrent prostate cancer within the prostatic fossa not treatable by surgery
* Non-regional lymphadenopathy (cM1a) or distant metastases (cM1b/c) as assessed by preoperative PSMA PET/CT.
* Castration resistance defined by clinical or biochemical progression despite a combined androgen blockade
* Known contraindications to hormone therapy, according to standard recommendations in force
* Patient with a psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule
* Ongoing androgen deprivation therapy (ADT) or within 6 months prior to surgery.
* Severe claustrophobia interfering with PET/CT scanning.
* Absence or withdrawal of an informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Clinical progression-free survival (CPFS) | 24 months
  CPFS is defined as time between randomization and the appearance of a recurrence (any N1 or M1) as suggested by PSMA PET/CT or symptoms related to progressive PC, or death due to any cause

SECONDARY OUTCOMES:
Metastasis-free survival (MFS) | 24 months
  Metastasis-free survival will be defined as the time between randomization and the appearance of a metastatic recurrence (any M1) as suggested by PSMA PET-CT.
Biochemical progression-free survival (BPFS) | 24 months
  Biochemical progression-free survival will be defined as the time between randomization and the development of biochemical progression ( three consecutive rises in prostate specific antigen (PSA) 1 week apart, resulting in two 50% increases over the nadir and PSA>2 ng/ml)
Castrate resistant prostate cancer (CRPC) | 10 years
  CRPC is defined as castrate serum testosterone<50 ng/dl plus biochemical progression, i.e., three consecutive rises in PSA 1 week apart, resulting in two 50% increases over the nadir and PSA>2 ng/ml.
Overall survival (OS) | 10 years
  Overall survival will be read as the time from trial randomization to the date of death from any cause
Incidence of adjuvant therapy | 10 years
  ADT, radiation therapy or additional salvage surgery
Patient reported QOL as per EORTC-QLQ C30 | 24 months
  Quality of life (QoL) will be assessed with the EORTC Core Quality of Life questionnaire's (QLQ-C30) global QoL scale ranging from 0 to 100, higher scores indicate better QoL
Patient reported QOL as per Expanded Prostate cancer Index Composite (EPIC) 26 | 24 months
  Quality of life (QoL) will be assessed with the EPIC 26 questionnaire, containing 26 items covering 5 domains: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better QOL.
Complications | 30 and 90 days
  Assessment of 99mTc-PSMA-I&S injection-related as well as surgery-related complication rate according to Clavien-Dindo.
Number of in-field recurrences | 24 months
  Recurrence measured by use of PSMA PET/CT in the template of 99mTc-PSMA-radioguided surgery (RGS) supported salvage surgery
Specificity of 99mTc-PSMA RGS for salvage surgery for recurrent PC compared to histologic evaluation | 30 days
  In percentage
Sensitivity of 99mTc-PSMA RGS for salvage surgery for recurrent PC compared to histologic evaluation | 30 days
  In percentage
Positive Predictive Value of 99mTc-PSMA RGS for salvage surgery for recurrent PC compared to histologic evaluation | 30 days
  In percentage
Negative Predictive Value of 99mTc-PSMA RGS for salvage surgery for recurrent PC compared to histologic evaluation | 30 days
  In percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek Hospital, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No